CLINICAL TRIAL: NCT00678873
Title: Single Incision Laparoscopic Cholecystectomy
Acronym: SILC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Homero Rivas, UT Southwestern
Organization: North Texas Veterans Healthcare System (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8843
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2008-08

CONDITIONS: Cholelithiasis
Keywords: Single Incision; Single Access; Surgery; Cholecystectomy
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy, Laparoscopic; Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical group (Experimental): Patients with ultrasound proven symptomatic cholelithiasis (gallstones).
  Interventions: Procedure: Single Incision Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Single Incision Laparoscopic Cholecystectomy — A single trans-umbilical incision laparoscopic cholecystectomy will be performed by standard fashion and under general anesthesia.
  Other Names: Single incision surgery; Single access surgery; Single incision laparoscopy; Single access laparoscopy; Laparoscopic cholecystectomy; Single access laparoscopic cholecystectomy; Cholecystectomy

SUMMARY:
The investigators aim to investigate the safety, feasibility and short-term outcomes of Single Incision Laparoscopic Cholecystectomy.

The investigators hypothesize that Single Incision Laparoscopic Cholecystectomy is safe and feasible.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the standard approach for the treatment of gallbladder disease. Laparoscopic cholecystectomy is now performed as an outpatient procedure and it commonly requires the use of 4 separate small incisions. Single incision or single access trans-umbilical surgery may provide less pain, scarring and may improve patient's overall satisfaction.

In this phase I trial we aim to evaluate the safety, feasibility and short-term outcomes of Single Incision Laparoscopic Cholecystectomy for the treatment of symptomatic cholelithiasis (gallstones).

ELIGIBILITY:
Inclusion Criteria:

* Adults male and female(>18 years old)
* Capable of giving informed consent
* Ultrasound proven cholelithiasis
* Symptomatic cholelithiasis
* Elective cholecystectomy

Exclusion Criteria:

* Pregnancy
* Contraindications for general anesthesia
* Morbid obesity
* Multiple previous abdominal surgeries
* Uncontrolled medical conditions
* Acute cholecystitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility | 12 months

SECONDARY OUTCOMES:
Short-term clinical outcomes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Homero Rivas, MD, Principal Investigator — UTSouthwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States